CLINICAL TRIAL: NCT02159365
Title: A Phase 2 Single Arm Study of Safety of Elotuzumab Administered Over Approximately 60 Minutes in Combination With Lenalidomide and Dexamethasone for Newly Diagnosed or Relapsed/Refractory Multiple Myeloma Patients
Brief Title: Study of Safety of Elotuzumab Administered Over Approximately 60 Minutes in Combination With Lenalidomide and Dexamethasone for Newly Diagnosed or Relapsed/Refractory Multiple Myeloma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA204-112
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Elotuzumab + Lenalidomide/Dexamethasone (Experimental): Elotuzumab 10 mg/kg solution intravenously weekly in cycle 1 and 2, then every other week, Lenalidomide 25 mg tablet by mouth Days 1-21 of each cycle / Dexamethasone 40 mg tablet by mouth / solution intravenously weekly until progression or discontinuation of Elotuzumab
  Interventions: Drug: Elotuzumab; Drug: Lenalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Elotuzumab
  Other Names: BMS-901608
Drug: Lenalidomide
  Other Names: Revlimid
Drug: Dexamethasone

SUMMARY:
To explore whether Elotuzumab dose administration over approximately 60 minutes is feasible and safe.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Documented evidence of active multiple myeloma:

  * Newly diagnosed, not candidate for transplant
  * Relapsed/refractory who have received up to 3 prior lines of therapy
* Prior Lenalidomide exposure is permitted only if the following criteria are fulfilled:

  * Not refractory to prior Lenalidomide which is defined as no progression while receiving Lenalidomide or within 60 days of last dose of Lenalidomide
  * Subject did not discontinue Lenalidomide due to a Grade ≥3 related adverse event (AE)

Exclusion Criteria:

* Target Disease Exceptions

  * Plasma cell leukemia
  * Monoclonal gammopathy of undetermined significance (MGUS)
  * Smoldering Myeloma
* Primary amyloidosis
* Polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2014-03-08 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2018-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (29):
- United States (29):
  - Acrc/Arizona Clinical Research Center, Inc., Tucson, Arizona
  - Highland Oncology Group, Fayetteville, Arkansas
  - Comprehensive Blood And Cancer Center, Bakersfield, California
  - California Cancer Associates for Research and Excellence, Encinitas, California
  - Compassionate Cancer Res Grp, Fountain Valley, California
  - Robert A. Moss, Md Facp, Inc., Fountain Valley, California
  - Loma Linda University Cancer Center, Loma Linda, California
  - Pacific Cancer Care, Monterey, California
  - Ventura County Hematology-Oncology Specialists, Oxnard, California
  - Wellness Oncology & Hematology, West Hills, California
  - James R. Berenson, MD, Inc., West Hollywood, California
  - Rocky Mountain Cancer Centers Llp, Denver, Colorado
  - Cancer Specialists Of North Florida, Jacksonville, Florida
  - Center For Cancer Care & Research, Lakeland, Florida
  - Baptist Health Medical Group Oncology, Miami, Florida
  - Oncology Specialists,S.C, Park Ridge, Illinois
  - Investigative Clinical Research Of Indiana, Llc, Indianapolis, Indiana
  - Horizon Oncology Research, Inc, Lafayette, Indiana
  - Clinical Research Alliance, Inc., New York, New York
  - St Francis Hospital, Greenville, South Carolina
  - Greenville Health System, Greenville, South Carolina
  - Texas Oncology, Dallas, Texas
  - Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Local Institution, Houston, Texas
  - Cancer Centers of South Texas, San Antonio, Texas
  - Blood & Cancer Center of East Texas, Tyler, Texas
  - Texas Oncology-McAllen South Second Street, Weslaco, Texas
  - Blue Ridge Cancer Care, Blacksburg, Virginia
  - Vista Oncology Inc., PS, Olympia, Washington

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 84 participants were enrolled. 70 participants were randomized and treated. Reasons for non-randomization/non-treatment were 10 no longer met study criteria, 1 withdrew consent, and 3 due to other reasons.
Groups:
- E-Ld: E-Ld refers to the combination of Elotuzumab with Lenalidomide/Dexamethasone.
Period: Overall Study
Arm/Group | E-Ld
Started | 70
Completed | 0 (Completed = Still on treatment)
Not Completed | 70
Not completed — Disease Progression | 23
Not completed — Other reasons | 11
Not completed — Administrative reason by Sponsor | 9
Not completed — Adverse Event unrelated to study drug | 9
Not completed — Study drug toxicity | 7
Not completed — Maximum clinical benefit | 3
Not completed — Subject request to discontinue treatment | 3
Not completed — Subject withdrew consent | 3
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: All Treated Participants
Arm/Group | E-Ld
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.40)
Age, Customized [Count of Participants; unit: Participants]
  < 75 years | 49
  >= 75 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 57
  Black or African American | 6
  Asian | 3
  American Indian or Alaska Native | 0
  Native Hawaiian or Other Pacific Islander | 0
  Other | 4
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — ECOG is a 6-item scale used to discern patient status by rating categories such as disease progression, daily functioning, appropriate treatment, and prognosis. Performance status is scored on a scale ranging from 0-5, with (best score) 0=fully active and able to carry on all pre-disease performance without restriction and (worst score) 5=death.
  Participants
    0 | 34
    1 | 32
    2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 3 or Grade 4 (G3/4) Infusion Reactions by the End of Treatment Cycle 2
Description: Infusion reaction was defined as any relevant sign or symptom occurring during or after elotuzumab infusion and considered by the investigator as an infusion reaction. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Potentially Life-threatening or disabling, Gr 5=Death.
Time Frame: From Day 1 to End of cycle 2 treatment (approximately 56 days)
Population: All Treated Participants
Measure: Number (95% Confidence Interval); unit: Participants
Arm/Group | E-Ld
Number analyzed (Participants) | 70
Participants | 0 [0 to 5.1]

2. Secondary Outcome: Number of Participants With Any Grade and Grade 3 or Grade 4 (G3/4) Infusion Reactions Over the Entire Study Period
Description: An infusion reaction in this study is defined as any relevant sign or symptom occurring during or after elotuzumab infusion and considered by the investigator as an infusion reaction. Grade (Gr) 1=Mild, Gr 2=Moderate, Gr 3=Severe, Gr 4=Potentially Life-threatening or disabling, Gr 5=Death.
Time Frame: Date of first dose up to 60 days post last dose (approximately 4 years)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | E-Ld
Number analyzed (Participants) | 70
Participants
  # of participants with any grade infusion reaction | 3
  # of participants with G3/4 infusion reaction | 1

ADVERSE EVENTS:
Time Frame: From Day 1 up to 60 days post last dose of study drug (approximately 4 years assessed up to July 2018)
Arm/Group | E-Ld
All-Cause Mortality (participants affected / at risk) | 8/70
Serious Adverse Events (participants affected / at risk) | 35/70
Other Adverse Events (participants affected / at risk) | 68/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld (N=70)
Anaemia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1
Atrial fibrillation (Cardiac disorders) | 5
Atrial flutter (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Visual impairment (Eye disorders) | 1
Colitis ischaemic (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Diverticular perforation (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Pyrexia (General disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Cavernous sinus thrombosis (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 5
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 2
Acute psychosis (Psychiatric disorders) | 1
Delirium (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E-Ld (N=70)
Anaemia (Blood and lymphatic system disorders) | 16
Neutropenia (Blood and lymphatic system disorders) | 13
Thrombocytopenia (Blood and lymphatic system disorders) | 8
Atrial fibrillation (Cardiac disorders) | 6
Dry eye (Eye disorders) | 4
Vision blurred (Eye disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 10
Constipation (Gastrointestinal disorders) | 20
Diarrhoea (Gastrointestinal disorders) | 26
Dry mouth (Gastrointestinal disorders) | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9
Nausea (Gastrointestinal disorders) | 19
Vomiting (Gastrointestinal disorders) | 8
Asthenia (General disorders) | 12
Chills (General disorders) | 7
Fatigue (General disorders) | 38
Influenza like illness (General disorders) | 4
Malaise (General disorders) | 4
Non-cardiac chest pain (General disorders) | 5
Oedema peripheral (General disorders) | 17
Pain (General disorders) | 4
Pyrexia (General disorders) | 15
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 10
Pneumonia (Infections and infestations) | 4
Sinusitis (Infections and infestations) | 5
Upper respiratory tract infection (Infections and infestations) | 24
Urinary tract infection (Infections and infestations) | 17
Fall (Injury, poisoning and procedural complications) | 8
Blood creatinine increased (Investigations) | 5
Vitamin d decreased (Investigations) | 7
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 9
Hyperglycaemia (Metabolism and nutrition disorders) | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 5
Hypokalaemia (Metabolism and nutrition disorders) | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 15
Back pain (Musculoskeletal and connective tissue disorders) | 17
Muscle spasms (Musculoskeletal and connective tissue disorders) | 20
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7
Myalgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Balance disorder (Nervous system disorders) | 4
Dizziness (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 13
Hypoaesthesia (Nervous system disorders) | 5
Neuropathy peripheral (Nervous system disorders) | 11
Peripheral sensory neuropathy (Nervous system disorders) | 4
Syncope (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 4
Anxiety (Psychiatric disorders) | 11
Insomnia (Psychiatric disorders) | 22
Dysuria (Renal and urinary disorders) | 5
Haematuria (Renal and urinary disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9
Night sweats (Skin and subcutaneous tissue disorders) | 7
Pruritus (Skin and subcutaneous tissue disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 13
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 5
Hypertension (Vascular disorders) | 4
Hypotension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.